CLINICAL TRIAL: NCT05089110
Title: Expression of Toll-like Receptors 3 , 7 and 9 in Peripheral Blood Mononuclear Cells of COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady Khalifa Musa Markos, Resident doctor, Assiut University
Other Study IDs: Immunity cells in COVID-19
Record Dates: First submitted 2021-10-21; First posted 2021-10-22 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: blood sample — 5 cm blood sample from COVID-19 patients

SUMMARY:
The aim of the study is to assess the expression of TLR 3, 7, and 9 in the population of peripheral blood mononuclear cells (PBMC) and in B lymphocytes (CD19+), T lymphocytes (CD4+ and CD8+) using flow cytometry in relation to the clinical parameters and outcome of COVID 19 patients .

DETAILED DESCRIPTION:
Abnormal stimulation of innate immunity may have a great influence on the immunopathogenesis of COVID 19 disease .The involvement of innate immunity receptors-toll-like receptors (TLR)-in the pathogenesis of COVID 19 is not adequately studied. The activation of these receptors by specific ligands is thought to initiate autoimmune processes[1]. TLR stimulation leads to increased expression of proinflammatory cytokines (IL-6, IFN

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old of both genders.
* Patients diagnosed as confirmed COVID-19 when they have a positive result of RT-PCR for SARS-CoV-2 RNA or confirmed diagnosis by typical clinical picture and radiological methods , according to the WHO and Egyptian Ministry of Health and Population (MOH) definitions, at Assiut University Hospital.

Exclusion Criteria:

* Children less than 18 years.
* Patients refusal to participate in the study

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as confirmed COVID-19 when they have a positive result of RT-PCR for SARS-CoV-2 RNA or confirmed diagnosis by typical clinical picture and radiological methods , according to the WHO and Egyptian Ministry of Health and Population (MOH) definitions, at Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Cytokines storm occurrence in COVID-19 patients | Baseline
  To assess whether the expression of toll-like receptors 3,7 and 9 in peripheral blood mononuclear cells related to the clinical status of COVID-19 patients and probability of cytokines storm occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Agamy, professor, Study Chair — Assiut University; Mohammad Adam, professor, Study Chair — Assiut University

REFERENCES:
- [Background] Matthay MA, Zemans RL, Zimmerman GA, Arabi YM, Beitler JR, Mercat A, Herridge M, Randolph AG, Calfee CS. Acute respiratory distress syndrome. Nat Rev Dis Primers. 2019 Mar 14;5(1):18. doi: 10.1038/s41572-019-0069-0. PMID 30872586
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578